CLINICAL TRIAL: NCT01763827
Title: A Double-blind, Randomized, Placebo and Ezetimibe-controlled, Multicenter Study to Evaluate Safety and Efficacy of Lipid Lowering Monotherapy With AMG 145 in Subjects With a 10-Year Framingham Risk Score of 10% or Less
Brief Title: Monoclonal Antibody Against PCSK9 to Reduce Elevated LDL-C in Subjects Currently Not Receiving Drug Therapy for Easing Lipid Levels-2
Acronym: MENDEL-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20110114
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Results first posted 2015-12-30 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Hyperlipidemia
Keywords: High cholesterol, Treatment for high cholesterol, Lowering cholesterol, Lowering high cholesterol, Hypercholesterolemia
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia | interventions — evolocumab; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo Q2W (Placebo Comparator): Participants received placebo subcutaneous injection once every 2 weeks (Q2W) and placebo tablets once a day for up to 12 weeks.
  Interventions: Biological: Placebo to Evolocumab; Other: Placebo to Ezetimibe
- Placebo QM (Placebo Comparator): Participants received placebo subcutaneous injection once every month (QM) and placebo tablets once a day for up to 12 weeks.
  Interventions: Biological: Placebo to Evolocumab; Other: Placebo to Ezetimibe
- Ezetimibe (Q2W) (Active Comparator): Participants received placebo subcutaneous injection once every 2 weeks and 10 mg ezetimibe orally once a day for up to 12 weeks.
  Interventions: Drug: Ezetimibe; Biological: Placebo to Evolocumab
- Ezetimibe (QM) (Active Comparator): Participants received placebo subcutaneous injection once a month and 10 mg ezetimibe orally once a day for up to 12 weeks.
  Interventions: Drug: Ezetimibe; Biological: Placebo to Evolocumab
- Evolocumab Q2W (Experimental): Participants received 140 mg evolocumab by subcutaneous injection once every 2 weeks and placebo tablets once a day for up to 12 weeks.
  Interventions: Biological: Evolocumab; Other: Placebo to Ezetimibe
- Evolocumab QM (Experimental): Participants received 420 mg evolocumab by subcutaneous injection once a month and placebo tablets once a day for up to 12 weeks.
  Interventions: Biological: Evolocumab; Other: Placebo to Ezetimibe

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha
  Arms: Evolocumab Q2W; Evolocumab QM
Drug: Ezetimibe — Administered orally once a day
  Other Names: Zetia
  Arms: Ezetimibe (Q2W); Ezetimibe (QM)
Biological: Placebo to Evolocumab — Administered by subcutaneous injection
  Arms: Ezetimibe (Q2W); Ezetimibe (QM); Placebo Q2W; Placebo QM
Other: Placebo to Ezetimibe — Administered orally once daily
  Arms: Evolocumab Q2W; Evolocumab QM; Placebo Q2W; Placebo QM

SUMMARY:
The primary objective was to evaluate the effect of 12 weeks of evolocumab subcutaneous (SC) monotherapy every 2 weeks (Q2W) and monthly (QM), compared with placebo and ezetimibe, on percent change from baseline in low-density lipoprotein cholesterol (LDL-C) in adults with a 10-year Framingham risk score of 10% or less.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 to ≤ 80 years of age
* National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III) Framingham risk score of 10% or less
* Fasting LDL-C ≥ 100 mg/dL (2.6 mmol/L) and <190 mg/dL
* Fasting triglycerides ≤ 400 mg/dL (4.5 mmol/L)

Exclusion Criteria:

* History of coronary heart disease
* New York Heart Association (NYHA) III or IV heart failure
* Uncontrolled cardiac arrhythmia
* Uncontrolled hypertension
* Diabetes mellitus (Type 1 diabetes, poorly controlled type 2 diabetes)
* Uncontrolled hypothyroidism or hyperthyroidism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2013-01-21 (Actual); Primary Completion 2013-10-10 (Actual); Study Completion 2013-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (75):
- United States (43):
  - Research Site, Birmingham, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Carmichael, California
  - Research Site, Encinitas, California
  - Research Site, San Diego, California
  - Research Site, Tustin, California
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Ponte Vedra, Florida
  - Research Site, Sanford, Florida
  - Research Site, Boise, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Bethesda, Maryland
  - Research Site, Brockton, Massachusetts
  - Research Site, Edina, Minnesota
  - Research Site, Olive Branch, Mississippi
  - Research Site, Las Vegas, Nevada
  - Research Site, Endwell, New York
  - Research Site, New Windsor, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Jackson, Tennessee
  - Research Site, Boerne, Texas
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Renton, Washington
  - Research Site, Seattle, Washington
- Australia (4):
  - Research Site, Darlinghurst, New South Wales
  - Research Site, Maroubra, New South Wales
  - Research Site, Carina Heights, Queensland
  - Research Site, Sherwood, Queensland
- Belgium (9):
  - Research Site, Anthée
  - Research Site, Brussels
  - Research Site, Gozée
  - Research Site, Gribomont
  - Research Site, Halen
  - Research Site, Ham
  - Research Site, Linkebeek
  - Research Site, Retie
  - Research Site, Tessenderlo
- Canada (4):
  - Research Site, Bay Roberts, Newfoundland and Labrador
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, Toronto, Ontario
  - Research Site, Granby, Quebec
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Ballerup Municipality
  - Research Site, Vejle
- France (2):
  - Research Site, Gières
  - Research Site, Grenoble
- South Africa (6):
  - Research Site, Alberton, Gauteng
  - Research Site, Johannesburg, Gauteng
  - Research Site, Parow, Western Cape
  - Research Site, Somerset West, Western Cape
  - Research Site, Worcester, Western Cape
  - Research Site, Bloemfontein
- Research Site, Seoul, South Korea
- Taiwan (2):
  - Research Site, Kaohsiung City
  - Research Site, Taipei
- Research Site, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Koren MJ, Lundqvist P, Bolognese M, Neutel JM, Monsalvo ML, Yang J, Kim JB, Scott R, Wasserman SM, Bays H; MENDEL-2 Investigators. Anti-PCSK9 monotherapy for hypercholesterolemia: the MENDEL-2 randomized, controlled phase III clinical trial of evolocumab. J Am Coll Cardiol. 2014 Jun 17;63(23):2531-2540. doi: 10.1016/j.jacc.2014.03.018. Epub 2014 Mar 29. PMID 24691094
- [Background] Daviglus ML, Ferdinand KC, Lopez JAG, Wu Y, Monsalvo ML, Rodriguez CJ. Effects of Evolocumab on Low-Density Lipoprotein Cholesterol, Non-High Density Lipoprotein Cholesterol, Apolipoprotein B, and Lipoprotein(a) by Race and Ethnicity: A Meta-Analysis of Individual Participant Data From Double-Blind and Open-Label Extension Studies. J Am Heart Assoc. 2021 Jan 5;10(1):e016839. doi: 10.1161/JAHA.120.016839. Epub 2020 Dec 16. PMID 33325247
- [Background] Koren MJ, Jones PH, Robinson JG, Sullivan D, Cho L, Hucko T, Lopez JAG, Fleishman AN, Somaratne R, Stroes E. A Comparison of Ezetimibe and Evolocumab for Atherogenic Lipid Reduction in Four Patient Populations: A Pooled Efficacy and Safety Analysis of Three Phase 3 Studies. Cardiol Ther. 2020 Dec;9(2):447-465. doi: 10.1007/s40119-020-00181-8. Epub 2020 Jun 20. PMID 32564340
- [Background] Kuchimanchi M, Grover A, Emery MG, Somaratne R, Wasserman SM, Gibbs JP, Doshi S. Population pharmacokinetics and exposure-response modeling and simulation for evolocumab in healthy volunteers and patients with hypercholesterolemia. J Pharmacokinet Pharmacodyn. 2018 Jun;45(3):505-522. doi: 10.1007/s10928-018-9592-y. Epub 2018 May 7. PMID 29736889
- [Background] Kasichayanula S, Grover A, Emery MG, Gibbs MA, Somaratne R, Wasserman SM, Gibbs JP. Clinical Pharmacokinetics and Pharmacodynamics of Evolocumab, a PCSK9 Inhibitor. Clin Pharmacokinet. 2018 Jul;57(7):769-779. doi: 10.1007/s40262-017-0620-7. PMID 29353350
- [Background] Shapiro MD, Minnier J, Tavori H, Kassahun H, Flower A, Somaratne R, Fazio S. Relationship Between Low-Density Lipoprotein Cholesterol and Lipoprotein(a) Lowering in Response to PCSK9 Inhibition With Evolocumab. J Am Heart Assoc. 2019 Feb 19;8(4):e010932. doi: 10.1161/JAHA.118.010932. PMID 30755061
- [Background] Stroes E, Robinson JG, Raal FJ, Dufour R, Sullivan D, Kassahun H, Ma Y, Wasserman SM, Koren MJ. Consistent LDL-C response with evolocumab among patient subgroups in PROFICIO: A pooled analysis of 3146 patients from phase 3 studies. Clin Cardiol. 2018 Oct;41(10):1328-1335. doi: 10.1002/clc.23049. Epub 2018 Oct 21. PMID 30120772
- [Background] Toth PP, Descamps O, Genest J, Sattar N, Preiss D, Dent R, Djedjos C, Wu Y, Geller M, Uhart M, Somaratne R, Wasserman SM; PROFICIO Investigators. Pooled Safety Analysis of Evolocumab in Over 6000 Patients From Double-Blind and Open-Label Extension Studies. Circulation. 2017 May 9;135(19):1819-1831. doi: 10.1161/CIRCULATIONAHA.116.025233. Epub 2017 Mar 1. PMID 28249876
- [Background] Toth PP, Jones SR, Monsalvo ML, Elliott-Davey M, Lopez JAG, Banach M. Effect of Evolocumab on Non-High-Density Lipoprotein Cholesterol, Apolipoprotein B, and Lipoprotein(a): A Pooled Analysis of Phase 2 and Phase 3 Studies. J Am Heart Assoc. 2020 Mar 3;9(5):e014129. doi: 10.1161/JAHA.119.014129. Epub 2020 Mar 2. PMID 32114889
- [Background] Wasserman SM, Sabatine MS, Koren MJ, Giugliano RP, Legg JC, Emery MG, Doshi S, Liu T, Somaratne R, Gibbs JP. Comparison of LDL-C Reduction Using Different Evolocumab Doses and Intervals: Biological Insights and Treatment Implications. J Cardiovasc Pharmacol Ther. 2018 Sep;23(5):423-432. doi: 10.1177/1074248418774043. Epub 2018 May 16. PMID 29768954
- [Background] May HT, Muhlestein JB, Ma Y, Lopez JAG, Coll B, Nelson J. Effects of Evolocumab on the ApoA1 Remnant Ratio: A Pooled Analysis of Phase 3 Studies. Cardiol Ther. 2019 Jun;8(1):91-102. doi: 10.1007/s40119-019-0133-6. Epub 2019 Mar 9. PMID 30852766
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men and women ≥ 18 to ≤ 80 years of age with fasting low-density lipoprotein cholesterol (LDL-C) ≥ 100 mg/dL and < 190 mg/dL and fasting triglycerides ≤ 400 mg/dL with a 10-year Framingham Risk Score of 10% or less were eligible for this study. The first participant was enrolled on 21 January 2013 and the last participant was enrolled 29 July 2013.
Pre-assignment Details: Participants received subcutaneous placebo corresponding to the once monthly dose volume during a 6 week screening period. Participants who completed the screening period and met final eligibility criteria were randomized 1:1:1:1:2:2 into 6 treatment groups. Randomization was stratified by LDL-C concentration (< 130 mg/dL or ≥ 30 mg/dL).
Period: Overall Study
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Started | 77 | 78 | 77 | 77 | 153 | 153
Received at Least 1 Dose of Study Drug | 76 | 78 | 77 | 77 | 153 | 153
Completed | 74 | 77 | 73 | 76 | 147 | 151
Not Completed | 3 | 1 | 4 | 1 | 6 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Decision by sponsor | 2 | 0 | 3 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM | Total
Number analyzed (Participants) | 77 | 78 | 77 | 77 | 153 | 153 | 615
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (10.3) | 52.6 (10.7) | 53.9 (11.3) | 53.0 (12.7) | 52.5 (13.7) | 52.9 (12.1) | 53.1 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 47 | 53 | 52 | 104 | 101 | 406
  Male | 28 | 31 | 24 | 25 | 49 | 52 | 209
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 2 | 3
  Asian | 9 | 8 | 7 | 10 | 12 | 12 | 58
  Black or African American | 4 | 6 | 6 | 6 | 9 | 9 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 64 | 63 | 63 | 60 | 132 | 129 | 511
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mixed Race | 0 | 0 | 1 | 0 | 0 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 6 | 8 | 9 | 11 | 14 | 21 | 69
  Not Hispanic or Latino | 71 | 70 | 68 | 66 | 139 | 132 | 546
Stratification Factor: Low-density Lipoprotein Cholesterol (LDL-C) [Number; unit: participants]
  < 130 mg/dL | 23 | 24 | 22 | 22 | 45 | 45 | 181
  ≥ 130 mg/dL | 54 | 54 | 55 | 55 | 108 | 108 | 434
LDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the full analysis set (all randomized participants who received at least 1 dose of investigational product (subcutaneously or orally).
  mg/dL | 139.5 (21.3) | 144.3 (23.9) | 143.3 (23.8) | 143.5 (23.1) | 141.7 (22.3) | 144.4 (23.3) | 142.9 (22.9)
Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the full analysis set
  mg/dL | 167.4 (25.8) | 172.8 (31.0) | 168.8 (28.9) | 169.4 (27.3) | 166.5 (25.6) | 170.4 (26.6) | 169.0 (27.2)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the full analysis set
  mg/dL | 103.7 (16.8) | 107.3 (19.9) | 107.2 (19.7) | 106.2 (17.8) | 104.5 (17.2) | 108.3 (17.9) | 106.2 (18.1)
Total Cholesterol/High-density Lipoprotein Cholesterol Ratio [Mean (Standard Deviation); unit: ratio] — Data are provided for the full analysis set
  ratio | 4.148 (1.311) | 4.444 (1.465) | 4.055 (1.082) | 4.335 (1.118) | 4.170 (1.170) | 4.175 (1.071) | 4.210 (1.191)
Apolipoprotein B/Apolipoprotein A-1 Ratio [Mean (Standard Deviation); unit: ratio] — Data are provided for the full analysis set
  ratio | 0.671 (0.193) | 0.713 (0.194) | 0.691 (0.187) | 0.712 (0.173) | 0.687 (0.169) | 0.707 (0.170) | 0.697 (0.178)
Lipoprotein(a) [Median (Inter-Quartile Range); unit: nmol/L] — Data are provided for the full analysis set
  nmol/L | 21.0 (62.9) [9.0 to 49.0] | 21.5 (84.0) [7.0 to 62.0] | 28.0 (79.1) [11.0 to 120.0] | 28.0 (65.7) [12.0 to 64.0] | 20.0 (61.5) [7.0 to 58.0] | 28.0 (86.9) [9.0 to 104.0] | 25.0 (74.5) [9.0 to 71.0]
Triglycerides [Median (Inter-Quartile Range); unit: mg/dL] — Data are provided for the full analysis set
  mg/dL | 113.5 (74.7) [83.3 to 178.0] | 118.0 (83.4) [85.5 to 178.5] | 112.5 (64.9) [83.5 to 158.0] | 116.5 (52.4) [90.0 to 159.0] | 112.0 (62.6) [81.5 to 147.5] | 119.0 (59.1) [82.5 to 168.5] | 115.3 (65.5) [83.5 to 163.0]
Very Low-density Lipoprotein Cholesterol (VLDL-C) Concentration [Median (Inter-Quartile Range); unit: mg/dL] — Data are provided for the full analysis set
  mg/dL | 22.5 (13.2) [16.8 to 34.3] | 23.8 (15.4) [17.0 to 35.5] | 22.5 (12.4) [16.5 to 32.0] | 23.5 (10.5) [18.0 to 31.5] | 22.5 (11.5) [16.5 to 29.5] | 23.5 (11.8) [16.5 to 33.5] | 23.0 (12.4) [16.5 to 32.5]
High-density Lipoprotein Cholesterol (HDL-C) Concentration [Median (Inter-Quartile Range); unit: mg/dL] — Data are provided for the full analysis set
  mg/dL | 57.0 (23.6) [43.8 to 77.3] | 54.0 (17.8) [44.5 to 65.5] | 58.5 (16.8) [47.0 to 69.5] | 53.5 (18.5) [42.0 to 67.5] | 53.0 (18.0) [44.5 to 67.0] | 56.5 (18.0) [46.5 to 65.5] | 55.3 (18.7) [44.5 to 67.5]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | 0.10 (1.67) | -1.34 (1.54) | -17.75 (1.67) | -18.57 (1.56) | -57.04 (1.23) | -56.12 (1.12)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; The null hypothesis was that there was no mean difference in the percent change from Baseline at Week 12 in LDL-C between evolocumab and placebo, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The model included treatment group, Baseline LDL-C level, scheduled visit and the interaction of treatment with scheduled visit; LS Mean Treatment Difference = -57.14, 95% CI 2-sided [-61.14 to -53.14], Standard Error of Mean 2.03 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The model includes treatment group, Baseline LDL-C level, scheduled visit and the interaction of treatment with scheduled visit; LS Mean Treatment Difference = -54.78, 95% CI 2-sided [-58.46 to -51.10], Standard Error of Mean 1.87 — Placebo is the reference
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; The null hypothesis was that there was no mean difference in the percent change from Baseline at Week 12 in LDL-C between evolocumab and ezetimibe, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -39.29, 95% CI 2-sided [-43.28 to -35.31], Standard Error of Mean 2.03 — Ezetimibe is the reference
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -37.55, 95% CI 2-sided [-41.24 to -33.86], Standard Error of Mean 1.88 — Ezetimibe is the reference

2. Primary Outcome: Percent Change From Baseline in LDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | -0.43 (1.45) | -1.41 (1.37) | -17.52 (1.46) | -19.12 (1.39) | -56.93 (1.07) | -58.81 (1.00)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; The null hypothesis was that there was no mean difference in the percent change from Baseline at the mean of Weeks 10 and 12 in LDL-C between evolocumab and placebo, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -56.50, 95% CI 2-sided [-59.95 to -53.04], Standard Error of Mean 1.76 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -57.40, 95% CI 2-sided [-60.66 to -54.14], Standard Error of Mean 1.66 — Placebo is the reference
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; The null hypothesis was that there was no mean difference in the percent change from Baseline at the mean of Weeks 10 and 12 in LDL-C between evolocumab and ezetimibe, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -39.41, 95% CI 2-sided [-42.87 to -35.94], Standard Error of Mean 1.76 — Ezetimibe is the reference
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -36.69, 95% CI 2-sided [-42.97 to -36.42], Standard Error of Mean 1.66 — Ezetimibe is the reference

3. Secondary Outcome: Change From Baseline in LDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
mg/dL | 1.2 (2.3) | 0.0 (2.1) | -23.1 (2.3) | -25.9 (2.1) | -78.4 (1.7) | -81.9 (1.5)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -79.6, 95% CI 2-sided [-85.0 to -74.2], Standard Error of Mean 2.7 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -81.9, 95% CI 2-sided [-87.0 to -76.9], Standard Error of Mean 2.6 — Placebo is the reference
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -55.3, 95% CI 2-sided [-60.7 to -49.9], Standard Error of Mean 2.7 — Ezetimibe is the reference
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -56.1, 95% CI 2-sided [-61.1 to -51.0], Standard Error of Mean 2.6 — Ezetimibe is the reference

4. Secondary Outcome: Change From Baseline in LDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
mg/dL | 1.9 (2.5) | -0.1 (2.4) | -23.4 (2.5) | -25.0 (2.4) | -78.4 (1.9) | -77.9 (1.7)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -80.4, 95% CI 2-sided [-86.4 to -74.3], Standard Error of Mean 3.1 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -77.8, 95% CI 2-sided [-83.4 to -72.2], Standard Error of Mean 2.8 — Placebo is the reference
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -55.0, 95% CI 2-sided [-61.1 to -49.0], Standard Error of Mean 3.1 — Ezetimibe was the reference
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The model includes treatment group, stratification factor, scheduled visit and the interaction of treatment with scheduled visit; LS Mean Treatment Difference = -52.9, 95% CI 2-sided [-58.5 to -47.3], Standard Error of Mean 2.9 — Ezetimibe was the reference

5. Secondary Outcome: Percentage of Participants Who Achieved a Mean LDL-C at Weeks 10 and 12 of Less Than 70 mg/dL
Time Frame: Weeks 10 and 12
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percentage of participants | 0.0 [0.0 to 4.8] | 0.0 [0.0 to 4.9] | 1.3 [0.2 to 7.2] | 2.8 [0.8 to 9.6] | 73.6 [65.7 to 80.2] | 71.3 [63.6 to 78.0]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Based on CMH test stratified by Baseline LDL-C level. For testing, non-achievement was imputed for participants with a missing value; Treatment Difference = 73.6, 95% CI 2-sided [64.4 to 80.2]
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 5, analysis 1]; Treatment Difference = 71.3, 95% CI 2-sided [62.2 to 78.0]
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 5, analysis 1]; Treatment Difference = 72.2, 95% CI 2-sided [62.4 to 78.9]
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 5, analysis 1]; Treatment Difference = 68.6, 95% CI 2-sided [58.3 to 75.5]

6. Secondary Outcome: Percentage of Participants Who Achieved LDL-C < 70 mg/dL at Week 12
Time Frame: Week 12
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percentage of participants | 1.4 [0.3 to 7.8] | 0.0 [0.0 to 5.2] | 1.4 [0.3 to 7.7] | 1.4 [0.3 to 7.8] | 72.9 [64.8 to 79.8] | 65.4 [57.1 to 72.9]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 5, analysis 1]; Treatment Difference = 71.5, 95% CI 2-sided [61.2 to 78.4]
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 5, analysis 1]; Treatment Difference = 65.4, 95% CI 2-sided [55.6 to 72.9]
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 5, analysis 1]; Treatment Difference = 71.5, 95% CI 2-sided [61.3 to 78.4]
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 5, analysis 1]; Treatment Difference = 64.0, 95% CI 2-sided [53.5 to 71.6]

7. Secondary Outcome: Percent Change From Baseline in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | -1.41 (1.34) | 1.32 (1.24) | -14.64 (1.35) | -16.48 (1.25) | -50.22 (0.99) | -51.96 (0.90)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -48.81, 95% CI 2-sided [-52.01 to -45.61], Standard Error of Mean 1.63 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -53.28, 95% CI 2-sided [-56.23 to -50.33], Standard Error of Mean 1.50 — Placebo is the reference
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -35.58, 95% CI 2-sided [-38.79 to -32.38], Standard Error of Mean 1.63 — Ezetimibe is the reference
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -35.49, 95% CI 2-sided [-38.44 to -32.53], Standard Error of Mean 1.50 — Ezetimibe is the reference

8. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | -0.31 (1.48) | 1.51 (1.38) | -14.89 (1.47) | -16.48 (1.39) | -50.12 (1.08) | -49.68 (1.01)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -49.81, 95% CI 2-sided [-53.34 to -46.27], Standard Error of Mean 1.79 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -51.19, 95% CI 2-sided [-54.49 to -47.90], Standard Error of Mean 1.67 — Placebo is the reference
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -35.23, 95% CI 2-sided [-38.74 to -31.71], Standard Error of Mean 1.78 — Ezetimibe is the reference
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -33.21, 95% CI 2-sided [-36.51 to -29.90], Standard Error of Mean 1.68 — Ezetimibe is the reference

9. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | 0.05 (1.51) | 1.54 (1.41) | -13.47 (1.52) | -14.75 (1.43) | -47.04 (1.12) | -49.39 (1.03)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -47.09, 95% CI 2-sided [-50.67 to -43.51], Standard Error of Mean 1.82 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -50.93, 95% CI 2-sided [-54.27 to -47.59], Standard Error of Mean 1.70 — Placebo is the reference
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -33.57, 95% CI 2-sided [-37.15 to -29.99], Standard Error of Mean 1.82 — Ezetimibe is the reference
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -34.64, 95% CI 2-sided [-37.99 to -31.28], Standard Error of Mean 1.71 — Ezetimibe is the reference

10. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | 0.59 (1.58) | 1.84 (1.53) | -13.17 (1.58) | -14.02 (1.54) | -47.21 (1.17) | -46.59 (1.12)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -47.81, 95% CI 2-sided [-51.56 to -44.05], Standard Error of Mean 1.91 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -48.43, 95% CI 2-sided [-52.07 to -44.79], Standard Error of Mean 1.85 — Placebo is the reference
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -34.04, 95% CI 2-sided [-37.78 to -30.30], Standard Error of Mean 1.90 — Ezetimibe is the reference
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -32.57, 95% CI 2-sided [-36.21 to -28.92], Standard Error of Mean 1.85 — Ezetimibe is the reference

11. Secondary Outcome: Percent Change From Baseline in Total Cholesterol/High Density Lipoprotein-cholesterol Ratio at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | 0.44 (1.29) | 6.42 (1.50) | -9.14 (1.29) | -11.90 (1.51) | -38.49 (0.95) | -39.41 (1.08)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -38.93, 95% CI 2-sided [-42.00 to -35.86], Standard Error of Mean 1.56 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -45.83, 95% CI 2-sided [-49.39 to -42.27], Standard Error of Mean 1.81 — Placebo is the reference
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -29.36, 95% CI 2-sided [-32.43 to -26.28], Standard Error of Mean 1.56 — Ezetimibe is the reference
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -27.51, 95% CI 2-sided [-31.08 to -23.94], Standard Error of Mean 1.81 — Ezetimibe is the reference

12. Secondary Outcome: Percent Change From Baseline in Total Cholesterol/High Density Lipoprotein-cholesterol Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | 1.18 (1.39) | 7.02 (1.67) | -10.03 (1.39) | -12.34 (1.68) | -38.45 (1.02) | -37.65 (1.21)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -39.63, 95% CI 2-sided [-42.97 to -36.30], Standard Error of Mean 1.69 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -44.67, 95% CI 2-sided [-48.66 to -40.68], Standard Error of Mean 2.03 — Placebo is the reference
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -28.42, 95% CI 2-sided [-31.73 to -25.10], Standard Error of Mean 1.68 — Ezetimibe is the reference
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -25.31, 95% CI 2-sided [-29.31 to -21.31], Standard Error of Mean 2.03 — Ezetimibe is the reference

13. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A1 Ratio at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | 1.01 (1.69) | 3.85 (1.77) | -13.39 (1.69) | -14.49 (1.79) | -48.12 (1.25) | -51.10 (1.29)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -49.12, 95% CI 2-sided [-53.12 to -45.12], Standard Error of Mean 2.03 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -54.95, 95% CI 2-sided [-59.12 to -50.78], Standard Error of Mean 2.12 — Placebo is the reference
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -34.73, 95% CI 2-sided [-38.73 to -30.73], Standard Error of Mean 2.03 — Ezetimibe is the reference
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -36.62, 95% CI 2-sided [-40.81 to -32.42], Standard Error of Mean 2.13 — Ezetimibe is the reference

14. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A1 Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | 1.12 (1.77) | 4.51 (1.90) | -12.69 (1.77) | -14.29 (1.92) | -48.45 (1.31) | -48.26 (1.39)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -49.57, 95% CI 2-sided [-53.78 to -45.36], Standard Error of Mean 2.14 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -52.77, 95% CI 2-sided [-57.28 to -48.26], Standard Error of Mean 2.29 — Placebo is the reference
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -35.76, 95% CI 2-sided [-39.95 to -31.57], Standard Error of Mean 2.13 — Ezetimibe is the reference
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 2]; LS Mean Treatment Difference = -33.97, 95% CI 2-sided [-38.48 to -29.45], Standard Error of Mean 2.29 — Ezetimibe is the reference

15. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | 0.12 (2.72) [-11.11 to 11.50] | 0.00 (2.96) [-11.82 to 8.33] | 0.00 (2.72) [-9.60 to 10.31] | -2.08 (3.01) [-18.18 to 5.56] | -18.37 (2.02) [-37.50 to 0.00] | -19.24 (2.17) [-38.80 to -4.79]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -18.48, 95% CI 2-sided [-25.28 to -11.68] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -19.24, 95% CI 2-sided [-23.20 to -15.28] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -18.37, 95% CI 2-sided [-24.39 to -12.35] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -17.15, 95% CI 2-sided [-23.23 to -11.08] — Median difference and 95% CI were obtained from McKean-Schrader algorithm

16. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | 0.00 (2.75) [-8.51 to 17.50] | 0.00 (3.26) [-10.53 to 8.11] | 0.00 (2.75) [-9.09 to 12.50] | -2.05 (3.28) [-17.19 to 8.33] | -20.41 (2.04) [-39.53 to 0.00] | -17.82 (2.39) [-38.46 to 0.00]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -20.41, 95% CI 2-sided [-27.76 to -13.06] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -17.82, 95% CI 2-sided [-24.51 to -11.12] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -20.41, 95% CI 2-sided [-28.13 to -12.69] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -15.77, 95% CI 2-sided [-24.39 to -7.14] — Median difference and 95% CI were obtained from McKean-Schrader algorithm

17. Secondary Outcome: Percent Change From Baseline in Triglycerides at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | -3.89 (3.64) [-18.85 to 11.24] | 4.89 (4.02) [-12.71 to 31.65] | -1.46 (3.60) [-15.03 to 18.41] | -3.97 (4.04) [-17.65 to 10.38] | -9.16 (2.65) [-24.19 to 11.03] | -15.71 (2.92) [-28.20 to 6.40]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.72, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -5.27, 95% CI 2-sided [-13.27 to 2.73] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -20.59, 95% CI 2-sided [-30.98 to -10.20] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.027, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -7.71, 95% CI 2-sided [-16.86 to 1.45] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p = 0.044, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -11.73, 95% CI 2-sided [-21.19 to -2.27] — Median difference and 95% CI were obtained from McKean-Schrader algorithm

18. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | -1.91 (3.13) [-18.58 to 11.46] | 2.01 (3.86) [-16.62 to 33.83] | 0.00 (3.15) [-13.26 to 17.54] | -2.41 (3.89) [-19.34 to 12.86] | -8.14 (2.31) [-26.14 to 10.13] | -15.64 (2.78) [-30.03 to 1.53]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.72, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -6.23, 95% CI 2-sided [-16.41 to 3.95] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -17.65, 95% CI 2-sided [-26.67 to -8.63] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.027, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -8.14, 95% CI 2-sided [-17.54 to 1.26] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p = 0.044, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -13.23, 95% CI 2-sided [-21.69 to -4.77] — Median difference and 95% CI were obtained from McKean-Schrader algorithm

19. Secondary Outcome: Percent Change From Baseline in Very Low Density Lipoprotein Cholesterol (VLDL-C) at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | -3.81 (3.09) [-19.16 to 9.97] | 4.22 (3.70) [-13.60 to 27.91] | -2.69 (3.12) [-16.54 to 16.67] | -3.33 (3.69) [-20.00 to 9.52] | -8.40 (2.28) [-25.43 to 10.91] | -16.17 (2.65) [-28.00 to 5.52]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.072, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -4.59, 95% CI 2-sided [-11.30 to 2.12] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -20.39, 95% CI 2-sided [-30.11 to -10.68] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.082, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -5.71, 95% CI 2-sided [-14.13 to 2.71] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p = 0.044, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baselie value; Median Treatment Difference = -12.84, 95% CI 2-sided [-22.14 to -3.54] — Median difference and 95% CI were obtained from McKean-Schrader algorithm

20. Secondary Outcome: Percent Change From Baseline in VLDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Ful analysis set
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | -1.58 (3.67) [-20.00 to 10.53] | 0.00 (3.93) [-16.67 to 33.33] | -0.94 (3.65) [-12.32 to 12.93] | -3.61 (3.87) [-19.23 to 14.29] | -9.52 (2.64) [-26.83 to 10.34] | -16.33 (2.80) [-30.73 to 2.51]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.72, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -7.94, 95% CI 2-sided [-18.81 to 2.92] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -16.33, 95% CI 2-sided [-25.64 to -7.02] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.082, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = -8.58, 95% CI 2-sided [-18.10 to 0.94] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p = 0.044, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The model includes treatment group, Baseline LDL-C level, scheduled visit and the interaction of treatment with scheduled visit as covariates; Median Treatment Difference = -12.72, 95% CI 2-sided [-20.89 to -4.54] — Median difference and 95% CI were obtained from McKean-Schrader algorithm

21. Secondary Outcome: Percent Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C) at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | -1.64 (1.26) [-8.41 to 5.03] | -4.67 (1.32) [-10.63 to -0.57] | -0.92 (1.27) [-10.11 to 7.29] | 0.00 (1.33) [-6.98 to 8.68] | 3.89 (0.93) [-1.35 to 11.55] | 3.81 (0.95) [-2.56 to 11.86]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.007, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = 5.53, 95% CI 2-sided [2.23 to 8.84] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = 8.48, 95% CI 2-sided [5.53 to 11.43] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.013, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = 4.81, 95% CI 2-sided [0.85 to 8.78] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p = 0.044, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline visit; Median Treatment Difference = 3.81, 95% CI 2-sided [-0.77 to 8.39] — Median difference and 95% CI were obtained from McKean-Schrader algorithm

22. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 76 | 78 | 77 | 77 | 153 | 153
percent change | -1.15 (1.43) [-9.09 to 6.06] | -5.27 (1.40) [-11.30 to 2.33] | -2.79 (1.42) [-8.57 to 8.74] | -1.47 (1.41) [-6.67 to 8.20] | 4.76 (1.05) [-2.86 to 12.82] | 4.06 (1.01) [-2.68 to 11.15]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.007, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = 5.91, 95% CI 2-sided [1.67 to 10.16] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = 9.33, 95% CI 2-sided [5.32 to 13.34] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 3: Comparison: Ezetimibe (Q2W) vs Evolocumab Q2W; Test type: Superiority or Other; p = 0.013, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = 7.56, 95% CI 2-sided [3.11 to 12.00] — Median difference and 95% CI were obtained from McKean-Schrader algorithm
Statistical Analysis 4: Comparison: Ezetimibe (QM) vs Evolocumab QM; Test type: Superiority or Other; p = 0.044, Quade test — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Adjusted for Baseline value; Median Treatment Difference = 5.53, 95% CI 2-sided [2.22 to 8.84] — Median difference and 95% CI were obtained from McKean-Schrader algorithm

ADVERSE EVENTS:
Time Frame: From the first dose of blinded investigational product until the end of the study (up to 14 weeks).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo Q2W | Placebo QM | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Serious Adverse Events (participants affected / at risk) | 0/76 | 1/78 | 0/77 | 1/77 | 3/153 | 1/153
Other Adverse Events (participants affected / at risk) | 9/76 | 4/78 | 10/77 | 4/77 | 12/153 | 12/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=76) | Placebo QM (N=78) | Ezetimibe (Q2W) (N=77) | Ezetimibe (QM) (N=77) | Evolocumab Q2W (N=153) | Evolocumab QM (N=153)
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=76) | Placebo QM (N=78) | Ezetimibe (Q2W) (N=77) | Ezetimibe (QM) (N=77) | Evolocumab Q2W (N=153) | Evolocumab QM (N=153)
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 2 | 1 | 4 | 5
Nasopharyngitis (Infections and infestations) | 1 | 2 | 4 | 2 | 3 | 3
Headache (Nervous system disorders) | 3 | 1 | 4 | 1 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.